CLINICAL TRIAL: NCT06728449
Title: Influence of Herbal Infusion of Cumin Seed, Ginger Root and Lemon Peel on Clinical Outcomes Among Patients With Hyperuricemia Associated Metabolic Syndrome
Brief Title: Influence of Herbal Infusion on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Maria Aslam, Maria Aslam, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-UOL-FAHS/808/2021
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: After the approval from the relevant authorities from The University of Lahore and Hospital, individuals meeting the ATP III criteria for metabolic syndrome (n = 330) will be selected for inclusion after taking consent. The selected participants will be randomly divided into control and 4 experimental groups. Anthropometric measurements, socio-economic status, nutrient intake and biochemical tests as fasting blood sugar level, triglyceride and cholesterol levels will be taken at beginning (0 day) and 60 days.
Who Masked: Participant, Care Provider
Masking Description: Double- Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Conventional therapy group (Active Comparator): Control group on Carbohydrate Controlled Diet with conventional therapy
  Interventions: Dietary Supplement: Conventional therapy
- Cumin tea group (Experimental): Intervention with Carbohydrate Controlled Diet along with Cumin Seeds Tea
  Interventions: Dietary Supplement: Cumin tea
- Ginger Tea Group (Experimental): Intervention with Carbohydrate Controlled Diet along with Ginger Tea
  Interventions: Dietary Supplement: Ginger Tea
- Lemon Peel Tea Group (Experimental): Intervention with Carbohydrate Controlled Diet along with Lemon Peel Tea
  Interventions: Dietary Supplement: Lemon Peel Tea
- Functional tea Group (Experimental): : Intervention with Carbohydrate Controlled Diet along with Functional Tea
  Interventions: Dietary Supplement: Functional Tea

INTERVENTIONS:
Dietary Supplement: Cumin tea — The preparation involved boiling 200 ml of water with 2 grams of cumin seeds. Patients were instructed to consume/ have tea twice a day i.e. in mid-morning and in the evening without sugar respectively.
  Arms: Cumin tea group
Dietary Supplement: Ginger Tea — The preparation involved boiling 200 ml of water with 2 grams of ginger. Patients were instructed to consume/ have tea twice a day i.e. in mid-morning and in the evening without sugar respectively.
  Arms: Ginger Tea Group
Dietary Supplement: Lemon Peel Tea — The preparation involved boiling 200 ml of water with 2 grams of lemon peel. Patients were instructed to consume/ have tea twice a day i.e. in mid-morning and in the evening without sugar respectively.
  Arms: Lemon Peel Tea Group
Dietary Supplement: Functional Tea — The preparation involved boiling 200 ml of water with 2 grams of functional tisane (0.6 g cumin seeds, 0.6 g ginger, and 0.6 g lemon peel) Patients were instructed to consume/ have tea twice a day i.e. in mid-morning and in the evening without sugar respectively.
  Arms: Functional tea Group
Dietary Supplement: Conventional therapy — A carbohydrate-controlled diet focuses on limiting refined carbohydrates and sugars and total carbohydrate restriction to 50-70gm per major meal.
  Arms: Conventional therapy group

SUMMARY:
After taking written informed consent patients, the selected participants were divided into control and experimental group randomly.

DETAILED DESCRIPTION:
Phase II: RCT Double- Blinded After the approval from the relevant authorities from The University of Lahore and Hospital, individuals meeting the ATP III criteria for metabolic syndrome (n = 330) will be selected for inclusion after taking consent. The selected participants will be randomly divided into control and experimental groups. Anthropometric measurements, socio-economic status, nutrient intake and biochemical tests as fasting blood sugar level, triglyceride and cholesterol levels were taken at beginning (0 day) and 60 days.

The study was conducted in three steps respectively I: Baseline Data II: Intervention III: Follow Up I: Baseline Data

Interview technique accompanied with questionnaire was used to get following information. Before intervention metabolic syndrome patients were assessed for:

Demographic Data:

The basic information based on demographic data such as age, gender, marital status, education, was taken.

A. Anthropometrics Height and Weight of the patients were measured in light clothing using stadiometer. Waist circumference were measured using a inches tape. Body mass index an indicator of nutritional status, is deliberated by individual's body weight in kg divided by the height in meter square (kg/m2)56.

B. Biochemical tests Blood pressure will be measured by a sphygmomanometer after a 15-minute rest in sitting position56.

Biomarkers (biochemical tests) as Fasting blood glucose (FBS), Lipid profile (total cholesterol, high density lipoprotein (HDL), Low Density Lipoprotein (LDL) and triglyceride levels), Liver functioning tests (LFT's) and Renal functioning tests were recorded.

Blood samples (10 mL) were taken after 12 to 14 hours of fasting state at the beginning and after 8 weeks of intervention. Fasting serum glucose, TG, TC, LDL-C, HDL, were determined .

Liver functioning tests Alanine transferase (ALT), Aspartate transferase (AST), and alkaline phosphatase (ALP) and kidney functioning tests were performed.

C. Clinical Findings The metabolic syndrome patients were assessed clinically to have an insight into nutritional deficiencies on the bases of sign and symptoms.

D. Dietary Recall/Data 24 hr recall and Food frequency checklist were used to assess the dietary intake of the patients II: Intervention T0: Control group on Carbohydrate Controlled Diet with conventional therapy T1: Intervention with Carbohydrate Controlled Diet along with Cumin Seeds Tea T2: Intervention with Carbohydrate Controlled Diet along with Ginger Tea T3: Intervention with Carbohydrate Controlled Diet along with Lemon Peel Tea T4: Intervention with Carbohydrate Controlled Diet along with Functional tea bags

Respondents / Metabolic syndrome patients were categorized into 5 groups and will be intervened for 2 months (60 days). Functional tea bags were given to patient and thereby instructed to consume/have tea twice a day i.e. in mid-morning and at evening without sugar and a standard cup size of 200 ml respectively.

The preparation involved boiling 200 ml of water with 2 grams of cumin seeds Patients were instructed to consume/ have tea twice a day i.e. in mid-morning and in the evening without sugar respectively.

III: Follow up During data collection the patient were informed to weekly on call follow up through their provided contact numbers. On call follow up were taken after every 2 weeks (15 days) to determine the Follow up/ dropout rate or any side effect being encountered by the patient. Patient were advised to visit the hospital after every fifteen days so that compliance was monitored and functional tea bags were given for respective days/ months and instance if there were any issue/ side effect that could be treated/ adjusted/ eliminated accordingly.

Reassessment:

After eight weeks Anthropometric and biochemical tests of patients will be taken to assess the result of intervention.

Data collection tool

* ATP III Criteria
* Questionnaire (Demographic profile)
* Food Frequency Checklist (FFQ)
* 24 hr Recall

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome patients either gender of 18 to 60 years will be included.
* Patients will be recruited on the basis of ATP III criteria
* Patients having any body mass index with confirmed diagnosis of Metabolic Syndrome and no use of any dietary supplement or no adherence to special diets at least one month prior to baseline

Exclusion Criteria:

Individuals with the following conditions will not be included as participants

* Genetically obese individuals
* Patients already on lipid lower drugs according to recommendation of physicians
* Patients taking any nutritional supplement
* Allergy to any drugs or specific foods
* Breastfeeding mothers
* Pregnant females
* Patients with any other medical history (renal diseases, infections, liver disorders, cardiovascular diseases)
* Patients receiving weight loss drugs or supplements, receiving any changes in diet or daily exercise programs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2021-03-07 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Waist Circumference | 60 days
  Normal range of waist circumference in men should be less than 40 inches and in women it should be less than 35 inches. Change in the waist circumference will be monitored during the trial.
  >102 cm ( >40 in ) >88 cm ( >35 in )
Serum Triglyceride Level | 60 days
  Change in serum Triglyceride Level were monitored before and after the trial
Serum HDL- Cholesterol Level | 60 days
  Change in Levels were monitored before and after the trial
Blood Pressure (Systolic and Diastolic) | 60 days
  Change in readings were monitored before and after the trial
Fasting Glucose Level | 60 days
  Change in readings were monitored before and after the trial

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aslam, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be shared in the form of research articles without the personal information of the participant

REFERENCES:
- [Background] Taghizadeh M, Memarzadeh MR, Abedi F, Sharifi N, Karamali F, Fakhrieh Kashan Z, Asemi Z. The Effect of Cumin cyminum L. Plus Lime Administration on Weight Loss and Metabolic Status in Overweight Subjects: A Randomized Double-Blind Placebo-Controlled Clinical Trial. Iran Red Crescent Med J. 2016 May 23;18(8):e34212. doi: 10.5812/ircmj.34212. eCollection 2016 Aug. PMID 27781121